CLINICAL TRIAL: NCT04345328
Title: Impact of the Bacterial Colonial Metabolism on Fecal Water Toxicity as Biomarkers of Future Colorectal Cancer Risk After Bariatric Surgery
Brief Title: Impact of Bariatric Surgery on the Gut Environment
Acronym: IMPORTUNE
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Full Professor at the Faculty of Medicine KU Leuven, KU Leuven
Other Study IDs: s59836
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric surgery; Toxicity; Colon; Microbial fermentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Feces Breath Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Roux-en-Y gastric bypass: Patients who were planned for surgery with Roux-en-Y gastric bypass and were operated
- Sleeve Gastrectomy: Patients who were planned for surgery with Sleeve Gastrectomy and were operated
- Control group: Obese patients involved in a weight loss program that focuses on diet and lifestyle changes

SUMMARY:
The purpose of this study is to investigate the impact of bariatric surgery on the gut health. Patients operated with Roux-en-Y gastric bypass or sleeve gastrectomy and obese patients who want too loose weight with a traditional weight-loss program, will be followed up for 1 year. In these patients, the investigators will measure toxicity parameters to understand better the health status of their colon after surgery. In a next phase, the measured toxicity will be linked with certain players that might cause this toxicity. Protein metabolites, formed from undigested protein by microbiota in the colon, are expected to be toxic agents for the colon. Therefore, the investigators will investigate the fate of ingested protein once the surgery patients are metabolically stabilized.

DETAILED DESCRIPTION:
To quantify protein assimilation after bariatric surgery, the investigators will perform in bariatric surgery patients (Roux-en- Y gastric bypass and Sleeve Gastrectomy) and in a control group a cross-sectional study with a single test day. On the test day, the study participants will consume a test meal that contains intrinsically labelled egg proteins and will take a capsule with 14C-glycocholic acid and a capsule with 3H-labelled polyethylene glycol. Participants will record a food diary 72h before and after the test day and during the test collect breath samples for 6h. Urine and stool will be collected respectively up to 24h and 72h after consumption of the test meal.

For the 1-year follow up study, the 3 patient groups (Roux-en-Y gastric bypass, Sleeve gastrectomy and control group with traditional weight loss therapy) will have 5 visits, a baseline visit and 4 visits after surgery or after starting traditional therapy. The time points after baseline include 2 weeks, 3 months, 6 months and 12 months. Each visit, a blood and stool sample will be collected, a 7-day food and stool diary will be registered and also weight loss will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Surgery patients (toxicity and protein assimilation) : BMI > 40 kg/m² or > 35 kg/m² if combined with either obstructive sleep apnoea syndrome, high blood pressure not controllable with 3 different medications or type II diabetes, (3) exclusion of other underlying causes of obesity by an endocrinologist, (4) having tried to lose weight on a non-surgical way for at least 1 year without result and (5) a positive advice from a multidisciplinary team consisting of a surgeon, endocrinologist, psychologist and dietitian.
* Obese control group in weight loss program (toxicity) : obese but otherwise healthy patients on a weight loss diet (BMI > 30 kg/m²) in the context of the weight-loss program organised at the Obesity Clinic of University Hospital Leuven.
* Control group (protein assimilation) : normal weight (BMI 25-30 kg/m²) or overweight (BMI 25-30 kg/m²).

Exclusion Criteria:

* Intake of antibiotics 1 months before the start of the study. Pre-and probiotics, laxatives and anti-diarrhea drugs 2 weeks before the start of the study.
* Surgery patients and control group (toxicity) : Gastrointestinal disease or major abdominal surgery in the past (except from appendectomy and cholecystectomy).
* Surgery patients and control group (protein assimilation) : Lung, liver, kidney and gastrointestinal disease or major abdominal surgery in the past (except from appendectomy, cholecystectomy and bariatric surgery). Vegan, vegetarian, lactose-or gluten-free diet. Pregnant or lactating women and subjects who participated in the last year in a study with irradiation exposure.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Surgery patient group was recruited at the University Hospital Leuven.
  * Obese control group was recruited at the Obesity Clinic of the University Hospital Leuven.
  * Normal and overweight control group was recruited among the employees and family members from employees of the University Hospital Leuven.
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in toxicity of faecal water up to 1 year after bariatric surgery | Baseline and 2 weeks, 3 months, 6 months and 1 year after surgery
  Faecal water toxicity : measured with a cell viability test. Toxicity : expressed as the dilution of faecal water at which 50 percent of the cells survive.
Degree of protein assimilation 6-24 months after bariatric surgery | 6-24 months after surgery
  Protein digestion, malabsorption and fermentation : assessed with stable isotope technology. Digestion and malabsorption : expressed as percent of the administered isotope dose. Fermentation : expressed as percent of maximal dose of the fermentation product that can be formed.

SECONDARY OUTCOMES:
Degree of fat malabsorption 6-24 months after bariatric surgery | 6-24 months after surgery
  Malabsorption of fat : calculated as ((fat intake- fat excretion)/fat intake)*100%, expressed as coefficient of fat absorption. Excretion : measured with the Van de Kamer method.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, PhD, Principal Investigator — KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Vlaams-Brabant, Belgium